CLINICAL TRIAL: NCT03216122
Title: Immediate vs Delayed Loading of Single Tooth Implants: Randomized Clinical Study
Brief Title: Immediate vs Delayed Loading of Single Tooth Implants
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Postgraduate Institute of Dental Sciences Rohtak (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Subramony perio
Record Dates: First submitted 2017-07-10; First posted 2017-07-13 (Actual); Last update posted 2021-12-17 (Actual); Status verified 2021-12

CONDITIONS: Implant Complication
MeSH Terms: interventions — Congresses as Topic; Immediate Dental Implant Loading

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control group (CG) (Active Comparator): The implant will be loaded after 3-4 months of placement (Conventional/Delayed Loading)
  Interventions: Procedure: Conventional/Delayed Loading
- Test group (TG) (Active Comparator): The implant will be loaded non-occlusally within 3-4 days of placement (Immediate Loading)
  Interventions: Procedure: Immediate Loading

INTERVENTIONS:
Procedure: Conventional/Delayed Loading
  Arms: Control group (CG)
Procedure: Immediate Loading
  Arms: Test group (TG)

SUMMARY:
Previous studies have shown high success rates of immediately loaded implants on par with conventionally loaded implants (DL), while a few studies have also reported failure rates. Various studies can be found in the English literature comparing IL to DL protocol, few of which used the flapless approach while few used cylindrical implants or were confined to maxillary anterior region. Furthermore, a perusal of literature revealed no study which used RVG for radiographic evaluation and evaluated the morbidity at the implant site in normal healthy adult population. Hence this study would help determine whether the IL protocol is on par with DL protocol, so as to reduce patient waiting time, prevent space closure and provide early patient satisfaction from an aesthetic stand point.

DETAILED DESCRIPTION:
Oral implants have become a reliable alternative to replace lost teeth as they have a very high survival rate. The survival rate of dental implants has improved significantly over the years and is often estimated to be above 90%. They support dental prosthesis, overdentures, crowns and bridges to restore oral function and aesthetics that the insertion of dental implants in bone has become one of the routine procedures in dental set up. It needs bone exposure which is associated with some amount of bone loss.

Osseointegrated implants are placed traditionally following a two stage protocol, wherein implants are left to heal unloaded for 3-4 months in mandible and 6-8 months in maxilla. Successful osseointegrated implants are anchored directly to bone. The presence of highly mineralized compact mature bone with many Haversian canals have been shown in the microscopy of retrieved implants from man and experimental animals. Regions of fibrous tissue interposition are not found. The newly formed bone has features of normality with marrow spaces filled with blood vessels.

However, in the presence of movement, a soft tissue interface may encapsulate the implant, causing its failure, that is, formation of a fibrous connective tissue rather than bone at the implant bone interface. A similar effect has been reported to occur in bone fractures that had been inadequately immobilized, resulting in a non-union of the fractured segments.

To minimize this, many clinicians advocate keeping the implants unloaded during the healing period. This traditional approach takes a longer treatment time and requires a second surgical intervention for connection of abutment to implant.

It would be beneficial to reduce the treatment period without affecting the success rate of the implants. Due to advancements in oral implantology, such as implant design and titanium surfaces treatment, the immediate loading concept has gained popularity by offering shortened treatment time, trauma reduction, decreased patient's anxiety, discomfort, improvement in function and esthetics. This treatment option also aims at maintenance of the hard and soft tissues and reducing the waiting period. Nowadays immediate and early loaded implants are becoming increasingly common due to the various benefits for patients.

Exact indication and considerations for the immediate loading protocol were defined for the first time in 2002 at the World Congress Consensus Meeting in Barcelona according to which adequate implant stability, controlled occlusal loads for full arch cases, non-occlusal loads for short span bridges and single teeth replacements are important considerations for a successful outcomes. According to this meeting, immediate functional (or occlusal) loading is defined in the treatment protocol, that is, when implants have been placed in the bone and have been restored with the use of restorations with occlusal contacts within 3-4 days of surgery, and immediate non-functional loading (IL) as restorations without occlusal contacts.

Occasionally immediately loaded implants have been associated with increased failure rates. it is therefore important to evaluate whether predictable results can be obtained according to the different loading protocols during replacement of a single tooth by implants.

The implant failure under immediate loading compared to delayed loading (DL) was evaluated in various randomized clinical trials. For the immediate loading group, the implant failure rate was 2.87% compared to 1.8% in the delayed loading group. Overall, there was no statistical significance in the difference in implant failure rate between these two groups.

Previous studies performed by Degidi et al. and Margossian et al. showed high success rates of immediately loaded implants placed in comparison with conventionally loaded implants. Recent studies performed by Merli et al and Romanos et al also proved that the success rate of the immediately loaded implants were on par, if not higher that the early or delayed loading protocols.

Various studies can be found in the English literature comparing IL to DL protocol, few of which used the flapless approach while few used cylindrical implants or were confined to maxillary anterior region. Furthermore, a perusal of literature revealed no study which used RVG for radiographic evaluation and evaluated the morbidity at the implant site in normal healthy adult population. Hence this study would help determine whether the IL protocol is on par with DL protocol, so as to reduce patient waiting time, prevent space closure and provide early patient satisfaction from an aesthetic stand point.

Therefore the purpose of the present study is to compare the results of immediate and delayed loading protocols. The null hypothesis is that there would be no difference in success rates, complications and peri-implant marginal bone level changes between the procedures, against the alternative hypothesis of a difference.

MATERIALS AND METHOD This study will be conducted in Department of Periodontics and Oral Implantology, Post Graduate Institute of Dental Sciences (PGIDS), Rohtak, Haryana.

STUDY POPULATION AND DESIGN A minimum of 24 individuals will be recruited from outpatient department of PGIDS, Rohtak and divided equally into test and control groups.

DISTRIBUTION OF SAMPLES Systemically healthy individuals will be divided randomly in two groups (control group & test group)

1. Control group (CG) - The implant will be loaded after 3-4 months of placement (Conventional/Delayed Loading)
2. Test group (TG) - The implant will be loaded non-occlusally within 3-4 days of placement (Immediate Loading)

Methodology The study will be conducted in two phases-

1. Pre surgical preparations:-which will include

   * Prior to implant preparation all patients will undergo a session of oral hygiene instructions and professionally delivered debridement procedures.
   * The patients will be subjected to complete hemogram analysis including platelet count, hemoglobin (Hb), bleeding time (BT), clotting time (CT), total leucocytes count (TLC), and differential leucocytes count (TLC).
2. Surgical preparations:-prior to surgery, 5% povidone iodine solution will be used for extra oral and intra oral asepsis.

Osteotomy procedure: - After administration of adequate amount of local anesthesia, a sharp full thickness incision will be given for elevation of a muco-periosteal flap at the middle of the crest followed by a crevicular incision on the adjacent teeth. After elevation of a full thickness flap, any sharp edges at the crest of the ridge will be smoothened. The crest should be at least 2mm wider than the diameter of the implant being used. The osteotomy site will be marked with a round bur and penetrate the cortex with a lanceolated drill. A 2mm twist drill will be used till the appropriate depth reference line- (drill speed 2000rpm). The orientation of the osteotomy can be checked using a direction indicator and taking an X-Ray/RVG with the indicator in place. Any changes in the direction, if required, can be made at this point. Sequentially the drills of increasing diameter will be used depending on the size of the implant selected observing anatomical landmarks (drill speed 800rpm). The final drill should be 0.5mm less than the implant diameter. Implant will be inserted by setting the torque 20-45Ncm, depending on the bone quality. Once the implant is fully seated, the implant driver will be pulled free from the implant connect the implant driver to the ratchet. X-ray/RVG will be taken to see the final position of the implant. Before adapting the soft tissue, the surgical site will be irrigated with normal saline to flush out any debris.

For the immediate loading (test) group, impression copings will be placed and impression made with addition silicone material and will be sent to lab for provisional restoration fabrication. The provisional restorations will be placed within 3-4 days of implant placement. The occlusal surface of the provisional restorations will be ground in order to avoid any contact with the opposite dentition in static and dynamic analysis. They will be recalled after 3-4 months for final prosthesis placement.

For the conventional loading (control) group, the flap will be sutured with a direct suture technique using 3-0 silk suture material. After one week patient will be recalled for suture removal. After three to four months of healing, radiographs will be taken to evaluate the mesial and distal crestal bone -implant interface before the abutment post is added to implant body. After this the cover screw will be removed after exposing it through the mucosa and low profile healing cap will be inserted. After 1-2 weeks of healing, the healing cap will be removed and transfer coping will be attached to implant. Impression will be made using Addition silicon impression material. Implant analogue will seated into coping in the impression and cast will be poured.

Impression and abutment will be sent to lab for fabrication of prosthesis. Prosthesis will be cemented using glass ionomer cement.

All the patients will be evaluated by Intra-oral radiographs and soft tissue parameters like Plaque Index, Gingival Index, Bleeding on Probing, Pocket Depth, Clinical Attachment Loss, Tooth mobility, Implant site morbidity. Data will be recorded at the time of implant placement and at 8 weeks, 4 months and 7 months of follow up primarily and total follow up period of 4 years.

Follow up and success criteria:- Assessments will be made at the time of placement of the implant (baseline), at 8 weeks, at 4 months and 7 months after placement of the implant and followed upto 4 years.

CLINICAL PARAMETERS based on 1st European Workshop on Periodontology

* For implant site and adjacent neighboring teeth site.
* Plaque index (PI) - SILNESS&LOE
* Bleeding on probing (BOP)
* Tooth mobility will be quantified by perio test
* Pocket probing depth (PPD)
* Clinical attachment level (CAL)
* Post-operative morbidity in terms of swelling, bruising, wound dehiscence, pus discharge will be observed clinically.
* Radiographic marginal bone loss/radiolucency will be observed by intraoral periapical x-ray/RVG using parallel cone technique and measured by Image J analysis.
* Periodontal probe (university of north carolina- UNC 15) probe will be used for recording periodontal parameters.

ELIGIBILITY:
Inclusion Criteria:

* • Patient having minimum single tooth edentulous space.

  * Adequate bone quality and quantity at the implant site.
  * Patient with acceptable oral hygiene (Plaque index<1.5).

Exclusion Criteria:

* • Medically compromised patient or patient taking immunosuppressive drugs or bisphosphonates which may complicate the treatment outcome.

  * Infection at the implant site and adjacent site.
  * History of bruxism or parafunctional habits.
  * Patient having history of bleeding disorder or on anticoagulant therapy.
  * Chronic smoker and using tobacco in any form.
  * Patients allergic to medication (Local anesthetic, Penicillin group of antibiotics, non- steroidal anti-inflammatory drugs) and implant.
  * Pregnant or lactating females.
  * Individuals with unacceptable oral hygiene (PI>1.5).
  * History of radiotherapy in the head and neck area

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2016-12-01 (Actual); Primary Completion 2018-04 (Actual); Study Completion 2021-10 (Actual)

PRIMARY OUTCOMES:
Crestal bone loss | 7 months primary, total time frame 4 years
  Interproximal marginal bone loss

CONTACTS AND LOCATIONS:
Overall Officials: SUBRAMONY BHAGAVATHEESWARAN, Principal Investigator — PGIDS ROHTAK
Locations (1):
- Post Graduate Institute of Dental Sciences, Rohtak, Haryana, India

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol